CLINICAL TRIAL: NCT00997724
Title: Feasibility of Assisted-VATS(Video-Assisted Thoracoscopic Surgery) Sleeve Lobectomy for Non-small Cell Lung Cancer
Brief Title: Assisted-VATS Sleeve Lobectomy for Non-small Cell Lung Cancer
Acronym: VATS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: The First Affiliated Hospital of Guangzhou Medical College, Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAHG96016
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: assisted-VATS (video-assisted thoracoscopic surgery); sleeve lobectomy; bronchoplasty
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- a-VATS (Experimental): Patients with NSCLC underwent assisted-VATS sleeve lobectomy with bronchoplasty.
  Interventions: Procedure: a-VATS

INTERVENTIONS:
Procedure: a-VATS — In brief, general anesthesia with selective lung ventilation was performed with the use of a double-lumen endotracheal tube. When postoperative mechanical ventilation was necessary, a standard endotracheal tube was substituted for the double-lumen tube. Patients were placed in the lateral decubitus position. Two thoracoports were placed in the sixth or seventh intercostal space (ICS) on the anterior axillary line and in the seventh or eighth ICS on the posterior axillary line; an anterolateral minithoracotomy (7 cm) was made in the fourth ICS for an upper lobectomy or in the fifth ICS for a middle or lower lobectomy.
  Other Names: assisted-VATS (video-assisted thoracoscopic surgery)

SUMMARY:
The purpose of this study is to examine the feasibility of assisted-VATS (video-assisted thoracoscopic surgery) sleeve lobectomy for non-small cell lung cancer for non-small cell lung cancer. Success is defined as assisted-VATS sleeve lobectomy without conversion. If success rate over 90%, assisted-VATS sleeve lobectomy is considered as feasible procedures for non-small cell lung cancer.

DETAILED DESCRIPTION:
Sleeve lobectomy is removal of a portion of a main stem bronchus in continuity with the adjacent lobe or bilobe followed by end-to-end bronchial anastomosis. The first reported bronchial sleeve resection was performed in 1947 at the Brompton Hospital in London, England, by Sir Clement Price Thomas. Whether sleeve resection is radical enough and indicated for patients who could tolerate pneumonectomy continues to be debated, although many recent reports have suggested that sleeve resection can achieve adequate curability rates. However, sleeve lobectomy has a definite role in the surgical management of lung cancer for patients whose pulmonary reserve is considered inadequate to permit pneumonectomy, and should be used anytime it is possible to achieve a margin-negative (R0) resection.

Although video-assisted thoracic surgery (VATS) is regarded as a minimally invasive procedure with good long-term survival results, many surgeons think that VATS is too complex and has too many technical limitations to be applied to bronchoplasty. Therefore, there are few reports in the literature of VATS bronchoplasty for lung cancer. The purpose of this study is to examine the feasibility of assisted-VATS (video-assisted thoracoscopic surgery) sleeve lobectomy for non-small cell lung cancer for non-small cell lung cancer. Success is defined as assisted-VATS sleeve lobectomy without conversion. If success rate over 90%, assisted-VATS sleeve lobectomy is considered as feasible procedures for non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (Squamous, adenosquamous, large cell, or poorly differentiated)
* Patients with central tumors located at the origin of a lobar bronchus.
* ECOG performance status 0-1
* Hematopoietic: WBC at least 4,000/mm^3; Platelet count at least 100,000/mm^3
* Hepatic: Bilirubin normal; AST/ALT no greater than 1.5 times upper limit of normal (ULN); Alkaline phosphatase no greater than 2.5 times ULN
* Renal: Creatinine clearance greater than 60 ml/min
* Cardiovascular: Cardiac function normal

Exclusion Criteria:

* Severe complications or infections
* Pregnant or breast-feeding women
* Clinically significant heart disease
* Uncontrolled hepatitis, chronic liver disease, or diabetes mellitus
* Another active cancer except properly treated carcinoma in situ of the cervix or basal/squamous cell skin carcinoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 1996-02; Primary Completion 2010-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
If success rate over 90%, assisted-VATS sleeve lobectomy is considered as feasible procedures for non-small cell lung cancer. (Success is defined as assisted-VATS sleeve lobectomy without conversion). | 3 months

SECONDARY OUTCOMES:
To evaluate the intraoperative(surgical duration, estimated blood loss), postoperative variables(mortality, morbidity, chest tube drainage duration, hospital stay), and 5-year survival rates. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD,FACS, Study Director — Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College
Locations (1):
- Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] He J, Shao W, Cao C, Yan TD, Wang D, Xiong X, Yin W, Xu X, Huang J. Long-term outcome of hybrid surgical approach of video-assisted minithoracotomy sleeve lobectomy for non-small-cell lung cancer. Surg Endosc. 2011 Aug;25(8):2509-15. doi: 10.1007/s00464-011-1576-6. Epub 2011 Feb 7. PMID 21298520